CLINICAL TRIAL: NCT04547465
Title: The Role of 2D Speckle-tracking Echocardiography in Diagnosis Chemotherapy-induced Cardiomyopathy in Breast Cancer Patients With High Cardiovascular Risk Factors
Brief Title: 2D Speckle-tracking Echocardiography in Chemotherapy-induced Cardiomyopathy With Cardiovascular Risk Factors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gia Dinh People Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 230/HĐĐĐ-ĐHYD
Record Dates: First submitted 2020-09-06; First posted 2020-09-14 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2022-08

CONDITIONS: Cardiomyopathy Due to Drug; Breast Cancer; Cardiovascular Risk Factor
MeSH Terms: conditions — Breast Neoplasms | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Echocardiography — 2D Speckle-tracking echocardiography

SUMMARY:
The aims of this study is to evaluate the role of 2D speckle-tracking echocardiography in diagnosis chemotherapy related left ventricular dysfunction in breast cancer patients with cardiovascular risks

DETAILED DESCRIPTION:
Chemotherapy induced cardiomyopathy is a serious adverse effect of anticancer treatments with poor long-term prognosis. In addition to the cumulative dose of anthracycline and trastuzumab, cardiovascular risks have been proven to be the "second hit" when dealing with chemotherapy related cardiomyopathy in breast cancer patients. Speckle-tracking echocardiography have had robust evidence in diagnosis the early stage of left ventricular dysfunction in various types of cancer treated by cardiotoxicity drugs. However, data is still lacking regarding the role of speckle-tracking echocardiography in breast cancer patients with cardiovascular risk

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients treated by anthracycline and/or trastuzumab
* Have at least one of these cardiovascular risks: age > 60, hypertension, atrial fibrillation, diabetes mellitus, dyslipidemia, chronic kidney disease, obesity, family history of cardiovascular diseases.

Exclusion Criteria:

* Left ventricular ejection fraction < 50% before chemotherapy
* Chronic heart failure with NYHA functional class >= II
* Significant valvular stenosis/regurgitation
* Acute heart failure due to acute coronary syndrome during follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients treated by anthracycline and/or trastuzumab with at least one of the cardiovascular risk factors
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-09-15 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of chemotherapy induced cardiomyopathy in breast cancer patients with cardiovascular risk | two year follow-up
  the incidence
The kinetics of left ventricular global longitudinal strain (LV-GLS) in breast cancer patients treated by anthracycline and/or trastuzumab | two year follow-up
  global longitudinal strain (percentage)
The cut-off value of global longitudinal strain (GLS) to predict chemotherapy induced cardiomyopathy in breast cancer patients treated by anthracycline and/or trastuzumab | two year follow-up
  global longitudinal strain (percentage)
The kinetics of right ventricular longitudinal strain (RV-GLS and RV-FWLS) in breast cancer patients treated by anthracycline and/or trastuzumab | two year follow-up
  longitudinal strain (percentage)
The kinetics of left atrial longitudinal strain (LASr, LAScd, LASct) in breast cancer patients treated by anthracycline and/or trastuzumab | two year follow-up
  longitudinal strain (percentage)

CONTACTS AND LOCATIONS:
Overall Officials: Hai H. Nguyen, Ph.D, Principal Investigator — Cardiology Department
Locations (1):
- Nguyen Hoang Hai, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided